CLINICAL TRIAL: NCT06563856
Title: A Phase 1, Open-Label, Single Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of TEPEZZA Subcutaneous Administration in Healthy Adult Subjects
Brief Title: A Study of TEPEZZA Subcutaneous Administration in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: HZNP-TEP-102
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Bioavailability; Bioequivalence
Keywords: Thyroid eye disease; Graves' ophthalmopathy; Graves' orbitopathy; Thyroid-associated ophthalmopathy; Immunology
MeSH Terms: conditions — Graves Ophthalmopathy | interventions — teprotumumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1: TEPEZZA Dose A SubQ (Experimental): Participants will receive Dose A of TEPEZZA administered SubQ.
  Interventions: Drug: TEPEZZA
- Cohort 2: TEPEZZA Dose B SubQ (Experimental): Participants will receive Dose B of TEPEZZA administered SubQ.
  Interventions: Drug: TEPEZZA
- Cohort 3: TEPEZZA Dose B Intravenously (IV) (Experimental): Participants will receive Dose B of TEPEZZA administered IV.
  Interventions: Drug: TEPEZZA
- Cohort 4: TEPEZZA Dose B and EDP SubQ (Experimental): Participants will receive coadministered doses of TEPEZZA Dose B and EDP SubQ.
  Interventions: Drug: TEPEZZA; Drug: EDP

INTERVENTIONS:
Drug: TEPEZZA — Administered as a SubQ injection or IV injection.
  Other Names: HZN-001
Drug: EDP — Administered as a SubQ injection.
  Arms: Cohort 4: TEPEZZA Dose B and EDP SubQ

SUMMARY:
The primary objective of this study is to assess the pharmacokinetics (PK) parameters of a single subcutaneous (SubQ) infusion of TEPEZZA with and without ENHANZE™ Drug Product (EDP) at 2 dose levels in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* The participant is able to provide written informed consent.
* The participant is male or female 18 to 55 years of age, inclusive.
* The participant has a body mass index (BMI) between 21 to 30 kg/m^², inclusive, and a minimum weight of 55 kg at Screening.
* The participant is considered by the investigator or designee to be in good general health as determined by medical history, clinical laboratory test results, vital sign measurements, 12-lead electrocardiogram (ECG) results, and physical examination findings at Screening.
* The participant has adequate venous access and can receive IV therapy.
* Female participants of childbearing potential must have a negative serum pregnancy test at Screening and Check-in and negative urine pregnancy tests at all other protocol-specified time points. Participants who are sexually active with a non-vasectomized male partner must agree to use 2 reliable forms of contraception during the study, one of which is recommended to be hormonal, such as an oral contraceptive.
* Female participants must agree not to donate an egg/oocyte from Day 1 until 180 days after receiving the study drug.

Male participants must agree not to donate sperm from Day 1 until 180 days after receiving the study drug.

-The participant is willing and able to comply with all protocol requirements and evaluations for the duration of the study.

Exclusion Criteria:

* The participant has a positive test result for hepatitis B surface antigen, hepatitis C virus (HCV) antibody, or human immunodeficiency virus (HIV) types 1 or 2 antibodies at Screening.
* The participant has a diagnosis of an autoimmune disease; or a history of HIV, hepatitis B virus (HBV), or HCV infection; a history of inflammatory bowel disease (IBD), or a history of or active thyroid eye disease (TED) at Screening.
* The participant has active liver disease or hepatic dysfunction at Screening or Check-in, as determined by alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels >1.5 times upper limit of normal (ULN).
* The participant has glycated hemoglobin (HbA1c) levels ≥8% and/or fasting glucose levels (after at least an 8-hour fast) >126 mg/dL (>7 mmol/L) at Screening.
* The participant has a seated resting blood pressure of <90/40 mmHg or >140/90 mmHg, or a seated pulse rate of <40 beats per minute (bpm) or >99 bpm or is considered clinically significant at Screening. One additional measurement can be taken if blood pressure and pulse rate are outside the specified limits.
* The participant has clinically significant 12-lead ECG abnormalities at Screening and Check-in or, in the opinion of the investigator, has a second- or third-degree atrioventricular (AV) block, or has any of the following:

QRS >120 msec

QT interval corrected for heart rate using Fridericia's formula (QTcF) >450 msec (males) or >470 msec (females)

PR interval >220 msec

* The participant has used any prescription (excluding hormonal birth control) or over-the-counter medications (except paracetamol [up to 2 g per day]), including herbal or nutritional supplements, within 14 days before receiving the study drug.
* The participant has a medical condition associated with an increased risk of bleeding - including a history of hematological diseases such as acquired platelet disorders; coagulation disorders - including drug-induced thrombocytopenia, idiopathic thrombocytopenia, or von Willebrand's Disease; or requires the use of antiplatelet or anticoagulant medication.
* Female participants who are lactating or planning to become pregnant from Screening through 180 days after receiving the study drug.
* Male participants who are planning to impregnate a female partner from Day 1 through 180 days after receiving the study drug.
* The participant has consumed alcohol-, caffeine-, or xanthine-containing products within 48 hours before the dose of study drug.
* The participant is a smoker or has used nicotine or nicotine-containing products (e.g., snuff, nicotine patch, nicotine chewing gum, mock cigarettes, or inhalers) within 3 months before receiving the study drug.
* The participant has a history of alcohol abuse or drug addiction within the past 6 months prior to Day 1 dosing.
* The participant has a positive test result for drugs of abuse, alcohol, or cotinine (indicating active current smoking) at Screening or before receiving the study drug.
* The participant is involved in strenuous activity or contact sports within 24 hours before receiving the study drug and during the study.
* The participant has donated blood, had significant blood loss, or received a transfusion of any blood or blood products within 60 days prior to Day 1 dosing or received a plasma donation within 7 days prior to Day 1 dosing.
* The participant has a history of relevant drug and/or food allergies (i.e., allergy or idiosyncratic reaction to components of TEPEZZA or excipients; prior hypersensitivity reactions to mAbs, EDP, or excipients; or any significant food allergy that could preclude a standard diet in the clinical unit).
* The participant participated in another investigational study within 30 days (or 5 half-lives of the study drug, whichever is longer) prior to dosing on Day 1. The 30-day window will be derived from the date of the last blood collection or dosing, whichever is later, in the previous study to the date of Day 1 of the current study.
* The participant has previously participated in a TEPEZZA investigational study or has received TEPEZZA or rHuPH20-containing products.
* The participant has received a COVID-19 vaccination within 6 weeks before receiving the study drug or during the study.
* The participant has a positive test for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). Note: Testing will be performed according to site procedures.
* The participant is mentally or legally incapacitated or has significant emotional problems at Screening or is expected to have them during the conduct of the study.
* The participant has a history or presence of a clinically significant medical or psychiatric condition or disease in the opinion of the investigator or designee.
* The participant had a history of any illness that, in the opinion of the investigator or designee, might confound the results of the study or pose an additional risk to the participant by participation in the study.
* In the opinion of the investigator or designee, the participant is not suitable for entry into the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2021-05-27 (Actual); Study Completion 2021-05-27 (Actual)

PRIMARY OUTCOMES:
Cohort 1, 2, and 4: Area Under the Serum Concentration-time Curve (AUC) From Time 0 Extrapolated to Infinity (AUCinf) of TEPEZZA | Day 1 pre-dose to Day 71
Cohort 1, 2, and 4: AUC From Time 0 to the Last Quantifiable Concentration (AUClast) of TEPEZZA | Day 1 pre-dose to Day 71
Cohort 1, 2, and 4: Percentage of the Area Extrapolated for Calculation of AUCinf (%AUCextrap) of TEPEZZA | Day 1 pre-dose to Day 71
Cohort 1, 2, and 4: Maximum Observed Serum Concentration (Cmax) of TEPEZZA | Day 1 pre-dose to Day 71
Cohort 1, 2, and 4: Last Quantifiable Serum Concentration (Clast) of TEPEZZA | Day 1 pre-dose to Day 71
Cohort 1, 2, and 4: Time to Maximum Observed Serum Concentration (Tmax) of TEPEZZA | Day 1 pre-dose to Day 71
Cohort 1, 2, and 4: Time of Last Quantifiable Serum Concentration (Tlast) of TEPEZZA | Day 1 pre-dose to Day 71
Cohort 1, 2, and 4: Apparent Terminal Elimination Rate Constant (λz) of TEPEZZA | Day 1 pre-dose to Day 71
Cohort 1, 2, and 4: Apparent Terminal Half-life (t1/2) of TEPEZZA | Day 1 pre-dose to Day 71
Cohort 1, 2, and 4: Apparent Serum Clearance (CL/F) of TEPEZZA | Day 1 pre-dose to Day 71
Cohort 1, 2, and 4: Apparent Volume of Distribution During the Terminal Phase (Vz/F) of TEPEZZA | Day 1 pre-dose to Day 71

SECONDARY OUTCOMES:
Cohort 3: AUCinf of TEPEZZA | Day 1 pre-dose to Day 71
Cohort 3: AUClast of TEPEZZA | Day 1 pre-dose to Day 71
Cohort 3: %AUCextrap of TEPEZZA | Day 1 pre-dose to Day 71
Cohort 3: Cmax of TEPEZZA | Day 1 pre-dose to Day 71
Cohort 3: Clast of TEPEZZA | Day 1 pre-dose to Day 71
Cohort 3: Tlast of TEPEZZA | Day 1 pre-dose to Day 71
Cohort 3: λz of TEPEZZA | Day 1 pre-dose to Day 71
Cohort 3: t1/2 of TEPEZZA | Day 1 pre-dose to Day 71
Cohort 3: Total Serum Clearance (CL) of TEPEZZA | Day 1 pre-dose to Day 71
Cohort 3: Estimated Volume of Distribution at Steady State (Vss) of TEPEZZA | Day 1 pre-dose to Day 71
Cohort 3: Volume of Distribution During the Terminal Phase (Vz) of TEPEZZA | Day 1 pre-dose to Day 71
Number of Participants Experiencing Treatment-emergent Adverse Events (TEAEs) | Up to approximately Day 71
  An adverse event (AE) is defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. Participants will be instructed to contact the investigator at any time after receiving the study drug, if any symptoms develop. A TEAE is defined as any event not present before exposure to study drug or any event already present that worsens in intensity or frequency after exposure.
Number of Participants Experiencing Serious Adverse Events (SAEs) | Up to approximately Day 71
  An AE is considered an SAE if, in the view of either the investigator or sponsor, it results in any of the following outcomes:
  * Death
  * Life-threatening AE
  * Inpatient hospitalization or prolongation of existing hospitalization
  * Persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
  * Congenital anomaly or birth defect.
Number of Participants with Detectable Anti-drug Antibodies (ADA) to TAPEZZA | Day 1 pre-dose to Day 71

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- PPD Development, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com